## MAKERERE UNIVERSITY COLLEGE OF HEALTH SCIENCES YALE UNIVERSITY

## VERBAL CONSENT TO PARTICIPATE IN A RESEARCH STUDY

| Hello, my name is | _ from Makerere University. I'd like to ask you to participate in a research |
|---|---|
| study about ways in which w | e can improve TB contact investigation. This is an important intervention |
| for finding undiagnosed peop | le with TB in the community. We are asking you to be in this study because |
| you will participate in quality | improvement meeting called a community of practice that will be taking |
| place at your clinic. We are in | nterested recording the meeting proceedings so that we can gain insign on |
| whether or not the meeting w | rere an implementation success. |
| meeting proceedings using a protected folder Box Secure. | ady, we every time you participate in these meetings we shall record all recorder at your facility and these will be transferred to a secure password Recordings will NOT be transcribed or translated. All recordings will be ving completion of the COP fidelity checklist. |
| All opinions shared during th | ese meetings in this will be kept confidential. Only key research staff will |
| listen to the recordings. Taki | ng part in this study is optional, and you can tell me if you want to stop |
| being in the study at any tim | e. Refusing to participate or ending your participation will not have any |
| effect on your employment | and any responses will be solely used for research purposes and not for |
| performance evaluation. | |
| Do you have any questions a | bout the study? |
| Would you like to participate | ? |
| If you have questions about number | this study in the future, you can contact the study coordinator at phone |